CLINICAL TRIAL: NCT02292355
Title: Effect of the Method Pilates in Women With Temporomandibular Disorders - Clinical Trial
Brief Title: Effect of the Method Pilates in Women With Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Jefferson Fagundes Loss, Doctor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URioGrande
Record Dates: First submitted 2014-11-06; First posted 2014-11-17 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Pain; Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders; posture; pain; clinical trial; Pilates
MeSH Terms: conditions — Pain; Temporomandibular Joint Disorders | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilates (Experimental): Intervention group will undergo Pilates sessions in addition to conventional treatment with occlusal splint
  Interventions: Other: Pilates
- Occlusal splint (No Intervention): Control group who receive conventional treatment with occlusal splint

INTERVENTIONS:
Other: Pilates — The intervention group will perform Pilates exercises for 15 weeks with frequency of twice weekly
  Other Names: Pilates exercises; Pilates method
  Arms: Pilates

SUMMARY:
Introduction: the influence of temporomandibular disorders (TMD) related to postural changes are yet no consensus, but it is believed that the imbalances of a system can influence another. Several techniques have been used to treat TMD and its associated problems, however there is a paucity of studies evaluating the effects of global treatments, such as Pilates, in individuals with TMD literature. Objective: To evaluate changes in the level of pain, the severity of TMD, the EMG activity of masticatory muscles and posture of young women undergoing training in Pilates, as well as correlating postural changes, pain level, severity of TMD and EMG activity of masticatory muscles. A randomized clinical trial with blinded assessors will be held. 40 patients divided randomly into two groups will be assessed, the control group (CG) who receive conventional treatment with occlusal splint and intervention group (IG), which in addition to conventional treatment will undergo Pilates sessions. Both groups will be formed for women aged 18 to 35 years with TMD and pain. The IG will receive treatment with the Pilates Method for 15 weeks with frequency of twice weekly and use occlusal splint as directed by the dentist. The CG will make use of occlusal splint alone. At the beginning and end of the 15 weeks the individuals are evaluated to verify the presence of TMD, TMD severity, pain, EMG evaluation of masticatory muscles and body posture. Data will be analyzed statistically.

DETAILED DESCRIPTION:
t-test or Mann-Whitney test will be used to compare data before and after 15 weeks of treatment.

Multiple Two-Way ANOVAs will be used to compare treatment and evaluation period, for each depended variable: effects of pain, severity of TMD, EMG activity of masticatory muscles and posture.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 35 years old;
* Possess temporomandibular disorder diagnosed by the Research Diagnostic Criteria for Temporomandibular Disorders (RDC / TMD) and classified into categories of severity of functional limitation through the Mandibular Function Impairment Questionnaire MFIQ
* Owning a complaint of pain in the TMJ region, classified as greater than 2.5 (moderate to high) by the Visual Analog Scale.

Exclusion Criteria:

* Have greater than 35 kg / m2 body mass index (BMI);
* Diagnosis of other disorders of the stomatognathic system;
* Have a history of any surgical procedure on the face, teeth and spine in the last six months;
* Possess severe pathologies of the spine (fractures, inflammatory diseases or tumors);
* Provide framework for intellectual disability or inability to give consistent information;
* Being in treatment for TMD, be it physical therapy, medical or dental care throughout the study period.
* Being practicing Pilates in the last six months;
* Being pregnant;
* Make use of dental prosthesis or appliance;
* Have a history of trauma to the face and temporomandibular joint in the last six months;
* Having presented temporomandibular joint dislocation in the last six months;
* Possess dental flaws between canines and molars.
* Provide cross bite, overbite or open bite;
* Presenting undershot or overshot jaw;
* Present vestibular disorders that may interfere with the balance
* Make use of continuous medication for pain or inflammation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2017-01-16 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measure | 15 weeks
  Pain intensity will be assessed using visual analog scale (VAS), which consists of a 10-cm horizontal line in which "0" means "No pain" and "10" means "The worst pain I can imagine".

SECONDARY OUTCOMES:
Severity of TMD | 15 weeks
  Severity of TMD will be assessed using the Mandibular Function Impairment Questionnaire (MFIQ).
EMG activity of masticatory muscles | 15 weeks
  EMG activity of masticatory muscles will be assessed using a surface eletromyography. Right and left masseter and temporalis muscles EMG activity will be record during 10 s of a masticatory activity
Posture | 15 weeks
  Women posture will be assessed with photogrametry

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson F Loss, Phd, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil